CLINICAL TRIAL: NCT02594228
Title: Effects of Increased Protein Intake and Exercise Training on Body Composition, Cardiovascular Health and Physical Performance
Brief Title: Protein Intake and Physical Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skidmore College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1012-227
Record Dates: First submitted 2015-10-29; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Physical Performance
MeSH Terms: interventions — Whey Proteins; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whey Protein and exercise training (Experimental): Six meals per day of 20 grams of protein, two of which were whey protein and 4 days per week of exercise training..
  Interventions: Behavioral: Whey Protein and exercise training
- Food Protein and exercise training (Experimental): Six meals per day of 20 grams of protein, all of which were whole food protein and 4 days per week of exercise training.
  Interventions: Behavioral: Food Protein and exercise training

INTERVENTIONS:
Behavioral: Whey Protein and exercise training — Six meals per day four of which were whole food and two of whey protein for an overall percentage of macronutrient intake of 25% protein and 4 days per week of exercise training
  Arms: Whey Protein and exercise training
Behavioral: Food Protein and exercise training — Six meals per day all of which were whole food protein for an overall percentage of macronutrient intake of 25% protein and 4 days per week of exercise training
  Arms: Food Protein and exercise training

SUMMARY:
A primary aim of the current proposal is to compare the effect of daily consumption of healthy lean protein as either whey protein (2 meals per day) or whole food (25% of total daily caloric intake) consumed as 6 small meals throughout the day, one of which is consumed immediately following exercise training (within 30 min) and another 2 hours prior to going to bed at night, over a 16 week period on muscle and fat mass, cardiovascular health, aerobic fitness, glucose, insulin, blood lipids, heart rate and muscle strength in overweight men and women.

DETAILED DESCRIPTION:
The primary purpose of this study is to examine the effects of increased healthy protein intake (25% of daily caloric intake as protein; 25% as healthy fats and oils; 50% as complex, unrefined carbohydrates) consumed as 6 small meals during the day in combination with exercise training 4 times per week, over a 16 week period in 25 overweight, but healthy males and females (30-60 yrs old). A secondary purpose is to compare the effects of consuming two of the 6 small meals during the day comprised of whole food protein source servings 20g/serving) with a matched group consuming whey protein for 2 daily protein servings (20g/serving). In the case of both groups, 1 serving will be consumed immediately following exercise [within 30 minutes] and 1 serving will be consumed 2 hours before going to bed. On non-exercise days, all participants will continue to consume 6 small meals per day in the same ratio of 25% lean protein, 25% healthy fats and oils, and 50% complex, unrefined carbohydrates but the groups will differ only in the composition of the last meal of the day consumed 2 hours before going to bed in which one group will consume protein (20g/serving) as whole food protein sources and the other group will consume a single serving of a whey protein supplement. The primary purpose of this study is to quantify changes in the following health outcomes at baseline and 16 weeks: total body muscle mass and fat mass (iDXA); abdominal fat mass (most highly related to cardiovascular and metabolic disease risk); blood sugar (glucose); blood lipids; insulin, aerobic fitness (assessed with a submaximal exercise test); and muscular strength (measured by 1 repetition maximum (RM) of the chest and leg press). The following additional measures will be assessed at baseline and 16 weeks: waist circumference; body weight, heart rate, blood pressure, and hunger (Visual Analog Scales).

ELIGIBILITY:
Inclusion Criteria:

* Each participant was screened prior to participating in the study using the Health and Fitness History, Physical Activity, and Physical Activity Readiness questionnaires administered by the investigators.
* Medical clearance was secured from the participant's primary care physician to verify no cardiovascular,metabolic or orthopedic issues that would prohibit them from performing the exercises for the duration of the study period
* Depending on the outcome of the health history, fitness and activity questionnaires and the physician's clearance, participants were informed of eligibility to participate in the study. A group meeting was scheduled for all eligible and interested participants to review the entire study. This process took place prior to administering any tests.

Exclusion Criteria:

* Participants were excluded if they smoked, had a whey protein intolerance, or orthopedic conditions that prohibited them from engaging in strenuous exercise

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Athletic Performance | baseline and post 16 week intervention
  Changes in one repetition maximum muscular strength of upper and lower body

SECONDARY OUTCOMES:
Total and Regional Body Composition | baseline and post 16 week intervention
  Changes in total and regional body fat assessed by dual energy xray

OTHER OUTCOMES:
Cardiometabolic Hormones | baseline and post 16 week intervention
  Changes in plasma insulin levels
Aerobic Fitness | baseline and post 12 week intervention
  Changes in oxygen consumption
Hunger Ratings | baseline and post 12 week intervention
  Changes in hunger visual analog scale ratings
Blood Lipids | baseline and post 12 week intervention
  Changes in total, LDL, HDL cholesterol
Blood Pressure | baseline and post 12 week intervention
  Changes in systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Paul j Arciero, Phd, Principal Investigator — Skidmore College